CLINICAL TRIAL: NCT06706128
Title: Reflex Rolling Versus Lung Squeezing Techniques On Pulmonary Functions In Premature Neonate With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pneumonia.
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): Consisted of twelve Preterm neonates
  Interventions: Other: reflex rolling technique
- Group (B) (Active Comparator): Consisted of twelve Preterm neonates
  Interventions: Other: lung squeezing technique

INTERVENTIONS:
Other: reflex rolling technique — received reflex rolling technique for 20 min, 5 days a week, for 2 weeks.
  Arms: Group (A)
Other: lung squeezing technique — lung squeezing technique for 20 min, 5 days a week, for 2 weeks
  Arms: Group (B)

SUMMARY:
Respiratory problems in neonates are one of the leading causes of neonatal morbidity and mortality in developing countries. These respiratory problems are seen in premature neonates, which mainly include respiratory distress syndrome (RDS), pneumonia, requiring ventilatory assistance or oxygen support

DETAILED DESCRIPTION:
The purpose of this study is to compare between the effect of reflex rolling and lung squeezing techniques on pulmonary functions in premature neonates with pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 1) Preterm neonates with pneumonia. 2) Neonates with 30-37 weeks of gestation admitted to NICU. 3) They were free from any major congenital malformation. 4) They were clinically and thermodynamically stable.

Exclusion Criteria:

* 1) Treatment with neurotropic drugs. 2) Interventricular hemorrhage. 3) Temperature >38 4) Respiratory and cardiac congenital anomalies. 5) Seizures. 6) Surgical procedures. 7) Genetic Disorders 8) Any segmental or lobar collapse confirmed on chest x-ray. 9) Major airway interventions including change of endo-tracheal tube, hand ventilation or bronchial lavage in the previous 12 hours.

Ages: 5 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | Respiratory Rate measured at day (0) at after 2 weeks
  Detected using monitors (Hunt Leigh Healthcare /United Kingdom).

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University for Science and Technology, Gamasa, Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: No